CLINICAL TRIAL: NCT03524521
Title: The Effect of Interval Training Using Body Weight on Body Composition in Sedentary Overweight and Obese Adults
Brief Title: Body Weight-Based Interval Training in Sedentary Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amanda R. Bonikowske, Senior Associate Consultant, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-010163
Record Dates: First submitted 2018-04-30; First posted 2018-05-14 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Body Weight Changes; Overweight and Obesity; Physical Activity
MeSH Terms: conditions — Body Weight Changes; Overweight; Obesity; Motor Activity | interventions — High-Intensity Interval Training; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Walking (Active Comparator): This arm is prescribed standard of care exercise prescription; 30 minutes of moderate intensity walking, 5 days/week.
  Interventions: Behavioral: Standard of Care
- Interval Training (Experimental): This arm is prescribed body-weight based interval training 3 days per week with progressive increase in exercise intervals and sets.
  Interventions: Behavioral: Interval Training

INTERVENTIONS:
Behavioral: Interval Training — Interval training is prescribed 3 days per week using 5 body weight exercises in a progressive fashion.
  Arms: Interval Training
Behavioral: Standard of Care — Walking prescribed to meet current exercise guidelines; 150 minutes per week.
  Arms: Standard Walking

SUMMARY:
Body-weight based interval training (IT) performed 3 times per week will lead to reductions in abdominal adiposity and reduce overall body fat percentage in overweight and obese sedentary adults more effectively than moderate intensity continuous training (MICT). Body-weight interval training will improve exercise capacity (peak VO2) in overweight/obese adults.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of the two home-based exercise groups.

The MICT group is the standard care group and will be instructed to walk for 30 minutes, 5 days per week at a moderate intensity. The goal is to accumulate 150 minutes of continuous aerobic exercise each week. Participants will be instructed on the use of the Rating of Perceived Exertion (RPE) scale during baseline testing and will be instructed to reach an RPE of 12-16. A heart rate monitor will be worn to monitor exercise intensity. Heart rate should reach ~70% of maximal heart rate.

The IT group will perform 5 body-weight exercises in three progressive phases. During the first 2 weeks the circuit will be completed twice, 30 second intervals, 90 seconds of rest. The exercises will be performed on 3 days of the week with at least one day of rest between exercise days (ideally Monday, Wednesday, Friday). The number of repetitions will increase to a maximum of 4 while the interval and rest periods increase to a maximum of 45 seconds each. The total time spent performing intervals by week 8 will be 15 minutes. A 2 minute warm up and 3 minute cool down will be performed, such as jumping jacks or simply walking. A heart rate monitor will be used to measure exercise intensity. Heart rate should reach approximately 90% of heart rate max during the intervals. Participants will be instructed on the use of the Rating of Perceived Exertion scale during baseline testing and will be instructed to reach an RPE of ≥17 during the high intensity intervals.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years of age
* Willing and able to provide informed consent
* Sedentary, overweight and obese adults (<90 minutes of moderate intensity exercise)
* BMI 25≤35
* Able to safely begin an exercise program
* Have a smartphone, and willing and able to download and use the Fitbit app

Exclusion Criteria:

* Unable to provide informed consent.
* Known cardiovascular disease, or uncontrolled hypertension,
* Diagnosed type 1 or 2 diabetes
* Women who are pregnant or plan to become pregnant in the next 3-4 months
* Orthopedic injury/limitation or any other contraindications to exercise.
* Medications that cause weight gain (steroids, HIV-related medications, etc.), or glucose lowering medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Change in Body fat percent | 12 weeks
  DEXA derived body fat %

SECONDARY OUTCOMES:
Change in Weight | 12 weeks
  Weight in kilograms
Change in peak VO2 | 12 weeks
  Peak VO2 in ml/kg/min
Visceral adipose tissue area | 12 weeks
  cm^2
Thigh adipose tissue area | 12 weeks
  cm^2

CONTACTS AND LOCATIONS:
Overall Officials: Amanda R Bonikowske, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials